CLINICAL TRIAL: NCT03777384
Title: EValuating the Safety Of De-escaLated Head and Neck Irradiation in HPV positivE Oropharynx Cancer in Non-smokers/Minimal Smokers
Status: Active, not recruiting | Type: Observational
Sponsor: Sanford Health (Other)
Responsible Party: Sponsor
Other Study IDs: SH EVOLVE
Record Dates: First submitted 2018-10-12; First posted 2018-12-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Oropharyngeal Cancer
Keywords: oropharynx; head and neck cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective, observational study evaluating the durability of local/regional control of previously published de-escalated radiotherapy protocols for patients with P16 positive oropharynx cancers who have minimal nicotine exposure who are not current uses (< 10 pack year smoking history; < 10 year history of any nicotine product [electronic cigarette, chewing tobacco]). Quality of Life measures will also be collected.

DETAILED DESCRIPTION:
This is a prospective, single-site, observational study in head and neck cancer participants. The purpose of this study is to provide a systematic platform to analyze, interpret, and track radiation dose de-escalation therapy and associated participant outcomes from treatments identified by these results.

Participants will be asked to complete quality of life questionnaires at regular time points before, during, and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologic confirmation of tumor of the oropharynx
* Radiation therapy (de-escalated head and neck irradiation) decision has been made
* Human Papilloma Virus (HPV) associated cancer as determined by positive p16 immunohistochemistry

  * HPV positivity is defined by p16 IHC staining of > 70% of tumor cells (strong and diffuse nuclear and cytoplasmic staining)
  * For cases that are indeterminate or if p16 testing cannot be accurately performed, HPV positivity can be confirmed by high-risk HPV DNA Testing which covers the following HPV subtypes: 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68
* < 10 pack year smoking history OR < 10 year nicotine use history
* No current tobacco/nicotine use (including electronic cigarettes and chewing tobacco)
* T1-T3, N0-N2 (AJCC8) requiring definitive therapy greater than surgery alone
* Ability to provide informed written consent
* Willingness to return to Sanford Cancer Center for follow-up
* Life expectancy > 12 weeks
* ECOG performance status < 3 (Appendix B)
* Adequate organ function for chemotherapy and radiotherapy

Exclusion Criteria:

* Any of the following because the inclusion criteria require delivery of radiotherapy and chemotherapy which is known to be genotoxic, and is associated with mutagenic and teratogenic effects: pregnant women, nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception.
* Prior head and neck radiotherapy
* Any factor precluding safe delivery of chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HPV positive oropharynx cancers who have minimal nicotine exposure who are not current uses (< 10 pack year smoking history; < 10 year history of any nicotine product [electronic cigarette, chewing tobacco]).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The durability of local disease control of de-escalated radiotherapy protocols in the community cancer center setting. | End of treatment to 5 years after end of treatment
  Number of participants who remain disease free from the end of treatment to 5 years after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Miran Blanchard, MD, Study Chair — Sanford Health
Locations (2):
- United States (2):
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Edith Cancer Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: No